CLINICAL TRIAL: NCT04725656
Title: Impact of the Nicotine Concentration on the Efficacy of a Nicotine Salt Vape Pod System as Smoking Cessation Tool
Brief Title: Concentration Impact Nicotine Salt
Acronym: CINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BASEC-ID: 2020-01875
Record Dates: First submitted 2021-01-13; First posted 2021-01-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation; Vaping
MeSH Terms: conditions — Smoking Cessation; Vaping

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active arm, low concentration (18 mg/mL) nicotine salt e-liquids (Active Comparator)
  Interventions: Procedure: Smoking cessation counseling; Other: Open system vape device and nicotine salt e-liquids
- Active arm, high concentration (59 mg/mL) nicotine salt e-liquids (Active Comparator)
  Interventions: Procedure: Smoking cessation counseling; Other: Open system vape device and nicotine salt e-liquids
- Control group (Other): Receive only smoking cessation counseling
  Interventions: Procedure: Smoking cessation counseling

INTERVENTIONS:
Procedure: Smoking cessation counseling — Smoking cessation counseling at baseline, week 1, and week 4.
Other: Open system vape device and nicotine salt e-liquids — Ad libitum use of nicotine salt e-liquids during three months.
  Arms: Active arm, high concentration (59 mg/mL) nicotine salt e-liquids; Active arm, low concentration (18 mg/mL) nicotine salt e-liquids

SUMMARY:
Double-blind (for the two active arms), randomized, three-arm (two active and one control) clinical trial investigating factors (e.g. nicotine concentration) influencing the success of smoking cessation strategies and possible health risks related to nicotine salt vaping.

DETAILED DESCRIPTION:
At the clinic screening visit demographics, smoking (including the Fagerström Test for Cigarette Dependence (FTCD) Questionnaire) and medical history, concomitant medication, vital signs, body mass index (BMI) and exhaled carbon monoxide (CO) will be assessed, and a physical examination will be performed. Saliva samples will be collected for cotinine and nicotine metabolite ratio (NMR) measurement, urine samples for urinary anabasine, 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), nicotine metabolites, tobacco-specific nitrosamines (TSNA), and VOC, and blood samples for genotyping, steroid levels, blood lipids, creatinine, and glucose.

After randomization the open system vape device and the nicotine salt e-liquids will be distributed to the participants of the two active arms. Use of e-liquids in the active arms will be ad libitum during three months and will be monitored by returned empty e-liquid bottles.

All groups will receive smoking cessation counseling at baseline, week 1, and week 4. Visits at the center at baseline, week 4, and 3 months will include questionnaires regarding TC and EC use, respiratory symptoms, liking, and adverse events, measurement of heart rate, blood pressure, BMI, blood steroid levels, HDL, LDL, creatinine and glucose, and measurement of urinary TSNA, VOC and nicotine metabolites. For participants self-reporting TC abstinence, exhaled CO validation and urinary anabasine and NNAL will be collected to verify tobacco abstinence.

A follow-up visit also assessing TC abstinence will take place at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) smokers (at least 5 TC per day for at least 12 months)
* Motivated to quit smoking as evidenced by signing the informed consent form at trial enrolment specifying that a target quit date will be set
* Exhaled CO ≥ 10 ppm or saliva cotinine of > 30 ng/ml (in case of borderline CO measurement of 6-10 ppm) at screening
* Willing to participate in the trial even if allocated to the control group
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study
* Signed informed consent form

Exclusion Criteria:

* Known hypersensitivity/allergy to a content of the e-liquid
* Pregnancy or breast feeding
* Intention to become pregnant during the course of the study
* Current regular use of EC or tobacco heating systems
* Use of NRT, varenicline, or bupropion in the month prior to the screening visit
* People who smoke tobacco combined with marijuana and do not currently want to quit marijuana use
* Participation in an interventional trial within 30 days prior to the screening visit
* Legal incapacity or limited legal capacity at screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence tobacco abstinence (in terms of non-inferiority) | 1 month
  Defined as no smoking, i.e. "not a puff", self-reported and confirmed by exhaled carbon monoxide (<10 ppm) and urinary anabasine levels (<3 ng/mL) when using low vs. high nicotine salt concentration e-liquids.
Volume of e-liquid used (in terms of superiority) | 1 month
  Volume of e-liquid used when using low vs. high nicotine salt concentration e-liquids.

SECONDARY OUTCOMES:
7-day point prevalence tobacco cigarette abstinence | 1 month
  Same as primary outcome using a less strict definition of tobacco cigarette abstinence, i.e. self-report of smoking no more than 5 cigarettes
Continuous tobacco cigarette abstinence | 1 month
  Self-reported continuous abstinence at 1 month (confirmed by exhaled carbon monoxide and urinary anabasine) using the stricter, i.e. "not a puff" and the less strict, i.e. "no more than 5 cigarettes" definition
7-day point prevalence tobacco cigarette abstinence | 3 and 6 months
  Self-reported 7-day point prevalence abstinence at 3 and 6 months (confirmed by exhaled carbon monoxide and urinary anabasine) using the stricter, i.e. "not a puff" and the less strict, i.e. "no more than 5 cigarettes" definition
Continuous tobacco cigarette abstinence | 3 and 6 months
  Self-reported continuous abstinence at 3 and 6 months (confirmed by exhaled carbon monoxide and urinary anabasine) using the stricter, i.e. "not a puff" and the less strict, i.e. "no more than 5 cigarettes" definition, and when allowing a 2-week "grace period" from the target quit date
Number of drop-outs | Through study completion
Time of dropping out | Through study completion
Urinary volatile organic compounds (VOC) | 1 and 3 months
  Change of non-nicotine toxicants (VOC) from baseline to 1 month and 3 months of nicotine salt use
Tobacco-specific nitrosamines (TSNA) | 1 and 3 months
  Change of non-nicotine toxicants (TSNA) from baseline to 1 month and 3 months of nicotine salt use
Liking/rating of trial product (active arms) | 1 and 3 months
  Questions regarding helpfulness in refraining from smoking, how satisfying and how good the e-cigarette tastes compared to the tobacco cigarettes, if they would recommend the assigned trial product to another smoker, and any potential practical problems they might have with the handling.
Respiratory symptoms | Up to 6 months
  Checklist with specific questions regarding shortness of breath, wheezing, cough or phlegm
Adverse events | Up to 6 months
  Checklist with specific questions regarding presence or absence of nausea, sleep disturbance, throat/mouth irritation or other
Total nicotine amount vaped | 1 and 3 months
Total volume of e-liquid consumed | 1 and 3 months
Steroid profiles | Baseline, 1, 3 and 6 months
  Steroid profiles in saliva, blood and urine
Number of cigarettes smoked per day among those who fail to quit | Through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Liakoni, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data that relates to individual, primary publications (and not the whole study database as such) will be deposited in the Bern Open Repository and Information System (BORIS). All efforts will be made to protect privacy and to de-identify the data. Data will be shared on request under the following conditions: A meaningful study question by the requester, outline of the planned analyses, valid methodology, signed data sharing agreement that contains a confidentiality agreement in case of sensitive data.